CLINICAL TRIAL: NCT06105138
Title: Exploring the Effects of Acute Cannabidiol Administration on Blood Alcohol Level and Intoxication in Adult Human Subjects
Brief Title: Cannabidiol Effects on Blood Alcohol Level and Intoxication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1903
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol; cannabidiol; craving
MeSH Terms: conditions — Alcoholism | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 200mg Cannabidiol (Experimental): - A single dose of 200mg commercially available (product code T-L-A-5) water-soluble solution supplied by Caliper Foods, to be consumed orally (mixed with water).
  Interventions: Dietary Supplement: 200mg Cannabidiol oral solution
- 30mg Cannabidiol, (Experimental): - A single dose of 30mg commercially available (product code T-L-A-5) water-soluble solution supplied by Caliper Foods, to be consumed orally (mixed with water).
  Interventions: Dietary Supplement: 30mg Cannabidiol oral solution
- Placebo (Placebo Comparator): - A single dose of water-soluble Placebo solution supplied by Caliper Foods, to be consumed orally (mixed with water).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 200mg Cannabidiol oral solution — 200mg cannabidiol administered in the laboratory prior to a standard dose of alcohol.
  The water-soluble product is standardized to 5.0% cannabidiol, 0.0% THC and composed of reverse-osmosis water, gum arabic, cannabidiol, MCT (Medium Chain Triglyceride) oil and citric acid. The same lot of Caliper water soluble CBD was used for both the 30 mg and 200 mg test variable. All CBD was sourced from the same lot of CDB isolate. The Caliper commercial product conforms to all standards set forth by the CDPHE (Colorado Dept of Public Health and Environment).
  Arms: 200mg Cannabidiol
Dietary Supplement: 30mg Cannabidiol oral solution — 30mg cannabidiol administered in the laboratory prior to a standard dose of alcohol.
  The water-soluble product is standardized to 5.0% cannabidiol, 0.0% THC and composed of reverse-osmosis water, gum arabic, cannabidiol, MCT (Medium Chain Triglyceride) oil and citric acid. The same lot of Caliper water soluble CBD was used for both the 30 mg and 200 mg test variable. All CBD was sourced from the same lot of CDB isolate. The Caliper commercial product conforms to all standards set forth by the CDPHE (Colorado Dept of Public Health and Environment).
  Arms: 30mg Cannabidiol,
Dietary Supplement: Placebo — Placebo administered in the laboratory prior to a standard dose of alcohol.
  The placebo was made up for the study and contained reverse-osmosis water, gum arabic, MCT (Medium Chain Triglyceride) oil, citric acid, plus the addition of a natural food color, used at <0.1%.
  Arms: Placebo

SUMMARY:
The main objectives of this study were to test if 2 different doses of Cannabidiol (compared to placebo) alter 1) breath alcohol concentration, 2) craving and subjective responses to alcohol or 3) cognitive performance following a standard dose of alcohol.

DETAILED DESCRIPTION:
Cannabidiol (CBD), is commonly found in the cannabis plant and has shown promise in treating alcohol use disorders (AUD). In this within-subjects, placebo-controlled, crossover study, the investigators explored the effects of two doses (200mg and 30mg) of plant-based CBD (compared to placebo CBD) on blood alcohol level, subjective effects of alcohol, craving and cognition over the course 4 hours after subjects consume a standardized dose of alcohol.

This pilot study was conducted at Colorado State University and volunteers were recruited from the local community. 36 individuals completed at least 1 study session and 22 completed all three sessions. At each session they received either placebo 30mg oral CBD or 200mg oral CBD prior to being given a standard dose of alcohol. They then remained in our laboratory for 4 hours and completed cognitive testing using the NIH toolbox Cognitive Battery, breath alcohol level measurements and self-reported intoxication ratings (using the The Biphasic Alcohol Effects Scale [BAES] and the The Subjective Effects of Alcohol Scale [SEAS]) and reported their craving levels using the Alcohol Urge Questionnaire (AUQ) every 30 minutes. They also provided 3 blood samples to measure blood-CBD levels at each session (prior to receiving the CBD, 25 minutes post-CBD ingestion and again 60 minutes later). Study sessions were separated by at least one week.

ELIGIBILITY:
Inclusion Criteria:

* 21-60 years old
* able to provide consent
* willing to consume CBD during the study
* report heavy drinking (>5 drinks [>4 for women] per occasion on at least 5 days/month in the past 3 months)
* not cannabis/CBD naive (i.e. THC or CBD use at least once in the past year), do not use cannabis regularly (i.e., less than monthly over past year), and no past-month cannabis use.

Exclusion Criteria:

* a regular or recent cannabis user (i.e. they used cannabis more often than monthly during the past year or used cannabis in the past month)
* were seeking treatment a substance use disorder (SUD) including AUD, taking medications to treat bipolar or psychotic disorders
* using nicotine every day
* taking blood thinning medications
* reported having a major medical condition contraindicating alcohol or CBD use (e.g., liver disease or heart disease)
* reported current suicidality
* met criteria for psychotic disorder, bipolar disorder or a current major depressive episode,
* reported using illicit drugs in the 30 days prior to beginning the study or tested positive for any illicit drugs
* were pregnant, breastfeeding or trying to become pregnant.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual (de-identified) participant data is to be made available to other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available upon request.

REFERENCES:
- [Result] Karoly HC, Drennan ML, Prince MA, Zulic L, Dooley G. Consuming oral cannabidiol prior to a standard alcohol dose has minimal effect on breath alcohol level and subjective effects of alcohol. Psychopharmacology (Berl). 2023 May;240(5):1119-1129. doi: 10.1007/s00213-023-06349-z. Epub 2023 Mar 20. PMID 36939855

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a crossover design. The total number of people enrolled was N=37. Of those 37, 1 was dropped from the study before completing any sessions, n=22 completed all three arms, n=4 completed only 2 appointments, and n=10 completed only 1 appointment.
Groups:
- 200mg Cannabidiol, 30mg Cannabidiol, Placebo: Experimental, 200mg CBD, 30mg CBD, Placebo
  Participants first received a single dose of 200mg CBD commercially available (product code T-L-A-5) water-soluble solution supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory. After a washout period of 7 days, they received a single dose of 30mg the same commercially available CBD product supplied by Caliper Foods, to be consumed orally (mixed with water) and administered in the laboratory. After a washout period of 7 days, they received a Placebo supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory.
  The water-soluble product is standardized to 5.0% cannabidiol, 0.0% THC and composed of reverse-osmosis water, gum arabic, cannabidiol, MCT (Medium Chain Triglyceride) oil and citric acid. The same lot of Caliper water soluble CBD was used for both the 30 mg and 200 mg test variable. All CBD was sourced from the same lot of CDB isolate. The placebo was made up for the study and contained reverse-osmosis water, gum arabic, MCT (Medium Chain Triglyceride) oil, citric acid, plus the addition of a natural food color, used at <0.1%. The Caliper commercial product conforms to all standards set forth by the CDPHE (Colorado Dept of Public Health and Environment).
- 200mg Cannabidiol, Placebo, 30mg Cannabidiol: Experimental, 200mg CBD, Placebo, 30mg CBD
  Participants first received a single dose of 200mg CBD commercially available (product code T-L-A-5) water-soluble solution supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory. After a washout period of 7 days, they received a Placebo supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory. After a washout period of 7 days, they received a single dose of 30mg the same commercially available CBD product supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory.
  The water-soluble product is standardized to 5.0% cannabidiol, 0.0% THC and composed of reverse-osmosis water, gum arabic, cannabidiol, MCT (Medium Chain Triglyceride) oil and citric acid. The same lot of Caliper water soluble CBD was used for both the 30 mg and 200 mg test variable. All CBD was sourced from the same lot of CDB isolate. The placebo was made up for the study and contained reverse-osmosis water, gum arabic, MCT (Medium Chain Triglyceride) oil, citric acid, plus the addition of a natural food color, used at <0.1%. The Caliper commercial product conforms to all standards set forth by the CDPHE (Colorado Dept of Public Health and Environment).
- 30mg Cannabidiol, Placebo, 200mg Cannabidiol: Experimental: 30mg CBD, Placebo, 200mg CBD
  Participants first received a single dose of 30mg CBD commercially available (product code T-L-A-5) water-soluble solution supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory. After a washout period of 7 days, they received a Placebo supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory. After a washout period of 7 days, they received a single dose of 200mg of the same commercially available CBD product supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory.
  The water-soluble product is standardized to 5.0% cannabidiol, 0.0% THC and composed of reverse-osmosis water, gum arabic, cannabidiol, MCT (Medium Chain Triglyceride) oil and citric acid. The same lot of Caliper water soluble CBD was used for both the 30 mg and 200 mg test variable. All CBD was sourced from the same lot of CDB isolate. The placebo was made up for the study and contained reverse-osmosis water, gum arabic, MCT (Medium Chain Triglyceride) oil, citric acid, plus the addition of a natural food color, used at <0.1%. The Caliper commercial product conforms to all standards set forth by the CDPHE (Colorado Dept of Public Health and Environment).
- 30mg Cannabidiol, 200mg Cannabidiol, Placebo: Experimental: 30mg CBD, 200mg CBD, Placebo,
  Participants first received a single dose of 30mg CBD commercially available (product code T-L-A-5) water-soluble solution supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory. After a washout period of 7 days, they received a single dose of 200mg of the same commercially available CBD product supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory. After a washout period of 7 days, they received a Placebo supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory.
  The water-soluble product is standardized to 5.0% cannabidiol, 0.0% THC and composed of reverse-osmosis water, gum arabic, cannabidiol, MCT (Medium Chain Triglyceride) oil and citric acid. The same lot of Caliper water soluble CBD was used for both the 30 mg and 200 mg test variable. All CBD was sourced from the same lot of CDB isolate. The placebo was made up for the study and contained reverse-osmosis water, gum arabic, MCT (Medium Chain Triglyceride) oil, citric acid, plus the addition of a natural food color, used at <0.1%. The Caliper commercial product conforms to all standards set forth by the CDPHE (Colorado Dept of Public Health and Environment).
- Placebo, 200mg Cannabidiol, 30mg Cannabidiol: Experimental: Placebo, 200mg CBD, 30mg CBD
  Participants first received a single dose of Placebo supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory. After a washout period of 7 days, they received a single dose of 200mg CBD commercially available (product code T-L-A-5) water-soluble solution supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory. After a washout period of 7 days, they received a single dose of 30mg of the same commercially available CBD product supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory.
  The water-soluble product is standardized to 5.0% cannabidiol, 0.0% THC and composed of reverse-osmosis water, gum arabic, cannabidiol, MCT (Medium Chain Triglyceride) oil and citric acid. The same lot of Caliper water soluble CBD was used for both the 30 mg and 200 mg test variable. All CBD was sourced from the same lot of CDB isolate. The placebo was made up for the study and contained reverse-osmosis water, gum arabic, MCT (Medium Chain Triglyceride) oil, citric acid, plus the addition of a natural food color, used at <0.1%. The Caliper commercial product conforms to all standards set forth by the CDPHE (Colorado Dept of Public Health and Environment).
- Placebo, 30mg Cannabidiol, 200mg Cannabidiol: Experimental: Placebo, 30mg CBD, 200mg CBD
  Participants first received a single dose of Placebo supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory. After a washout period of 7 days, they received a single dose of 30mg CBD commercially available (product code T-L-A-5) water-soluble solution supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory. After a washout period of 7 days, they received a single dose of 200mg of the same commercially available CBD product supplied by Caliper Foods, to be consumed orally (mixed with water), and administered in the laboratory.
  The water-soluble product is standardized to 5.0% cannabidiol, 0.0% THC and composed of reverse-osmosis water, gum arabic, cannabidiol, MCT (Medium Chain Triglyceride) oil and citric acid. The same lot of Caliper water soluble CBD was used for both the 30 mg and 200 mg test variable. All CBD was sourced from the same lot of CDB isolate. The placebo was made up for the study and contained reverse-osmosis water, gum arabic, MCT (Medium Chain Triglyceride) oil, citric acid, plus the addition of a natural food color, used at <0.1%. The Caliper commercial product conforms to all standards set forth by the CDPHE (Colorado Dept of Public Health and Environment).
Period: Overall Study
Arm/Group | 200mg Cannabidiol, 30mg Cannabidiol, Placebo | 200mg Cannabidiol, Placebo, 30mg Cannabidiol | 30mg Cannabidiol, Placebo, 200mg Cannabidiol | 30mg Cannabidiol, 200mg Cannabidiol, Placebo | Placebo, 200mg Cannabidiol, 30mg Cannabidiol | Placebo, 30mg Cannabidiol, 200mg Cannabidiol
Started | 6 | 4 | 4 | 7 | 12 | 3
Completed | 3 | 3 | 0 | 5 | 8 | 3
Not Completed | 3 | 1 | 4 | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Population: All 36 individuals who participated in the study (i.e., who completed at least one study session) were included in baseline descriptive analyses
Groups:
- Entire Sample: Individuals (N=36) who completed at least 1 session
Arm/Group | Entire Sample
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 17
Race/Ethnicity, Customized [Number; unit: participants]
  White | 34
  Mixed Race | 1
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 36
Alcohol Use Disorders Identification Test [Mean (Standard Deviation); unit: units on a scale] — Alcohol Use Disorders Identification Test, which measures the severity of alcohol use problems and indicates the likelihood that someone is experiencing hazardous alcohol use.
  Total score ranges from 0-40 (where higher values represent more problems with alcohol and a higher likelihood of hazardous alcohol use)
  units on a scale | 9.7 (4.7)
Beck Depression Inventory [Mean (Standard Deviation); unit: units on a scale] — Beck Depression Inventory, which measures current depression symptoms. The range of possible total scores is 0 to 63, where higher scores indicate more severe depression.
  units on a scale | 7.3 (6.3)
Beck Anxiety Inventory [Mean (Standard Deviation); unit: units on a scale] — Beck anxiety inventory, which measures current anxiety symptoms. Total score ranges from 0 to 63, with higher scores indicating greater severity of anxiety.
  units on a scale | 4.4 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Breath Alcohol Concentration (BrAC)
Description: Breath alcohol level will be measured using a breathalyzer repeatedly during the experimental session
Time Frame: Timepoint 1 (20 minutes after alcohol consumption is complete)
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- 200mg Cannabidiol: - A single dose of 200mg commercially available (product code T-L-A-5) water-soluble solution supplied by Caliper Foods, to be consumed orally (mixed with water).
  200mg Cannabidiol oral solution: 200mg cannabidiol administered in the laboratory prior to a standard dose of alcohol.
  The water-soluble product is standardized to 5.0% cannabidiol, 0.0% THC and composed of reverse-osmosis water, gum arabic, cannabidiol, MCT (Medium Chain Triglyceride) oil and citric acid. The same lot of Caliper water soluble CBD was used for both the 30 mg and 200 mg test variable. All CBD was sourced from the same lot of CDB isolate. The Caliper commercial product conforms to all standards set forth by the CDPHE (Colorado Dept of Public Health and Environment).
- 30mg Cannabidiol,: - A single dose of 30mg commercially available (product code T-L-A-5) water-soluble solution supplied by Caliper Foods, to be consumed orally (mixed with water).
  30mg Cannabidiol oral solution: 30mg cannabidiol administered in the laboratory prior to a standard dose of alcohol.
  The water-soluble product is standardized to 5.0% cannabidiol, 0.0% THC and composed of reverse-osmosis water, gum arabic, cannabidiol, MCT (Medium Chain Triglyceride) oil and citric acid. The same lot of Caliper water soluble CBD was used for both the 30 mg and 200 mg test variable. All CBD was sourced from the same lot of CDB isolate. The Caliper commercial product conforms to all standards set forth by the CDPHE (Colorado Dept of Public Health and Environment).
- Placebo: - A single dose of water-soluble Placebo solution supplied by Caliper Foods, to be consumed orally (mixed with water).
  Placebo: Placebo administered in the laboratory prior to a standard dose of alcohol.
  The placebo was made up for the study and contained reverse-osmosis water, gum arabic, MCT (Medium Chain Triglyceride) oil, citric acid, plus the addition of a natural food color, used at <0.1%.
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
g/dL | 0.065 (0.017) | .067 (.015) | .070 (.014)

2. Primary Outcome: Breath Alcohol Concentration (BrAC)
Description: Breath alcohol level will be measured using a breathalyzer repeatedly during the experimental session
Time Frame: Timepoint 2 (30 minutes after Timepoint 1)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
g/dL | 0.066 (0.014) | 0.067 (0.013) | 0.069 (0.011)

3. Primary Outcome: Breath Alcohol Concentration (BrAC)
Description: Breath alcohol level will be measured using a breathalyzer repeatedly during the experimental session
Time Frame: Timepoint 3 (30 minutes after Timepoint 2)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
g/dL | 0.059 (0.011) | 0.058 (0.010) | 0.061 (0.008)

4. Primary Outcome: Breath Alcohol Concentration (BrAC)
Description: Breath alcohol level will be measured using a breathalyzer repeatedly during the experimental session
Time Frame: Timepoint 4 (30 minutes after Timepoint 3)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
g/dL | 0.048 (0.010) | 0.049 (0.009) | 0.050 (0.008)

5. Primary Outcome: Breath Alcohol Concentration (BrAC)
Description: Breath alcohol level will be measured using a breathalyzer repeatedly during the experimental session
Time Frame: Timepoint 5 (30 minutes after Timepoint 4)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
g/dL | .040 (.009) | .040 (.009) | .041 (.007)

6. Primary Outcome: Breath Alcohol Concentration (BrAC)
Description: Breath alcohol level will be measured using a breathalyzer repeatedly during the experimental session
Time Frame: Timepoint 6 (30 minutes after Timepoint 6)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
g/dL | 0.032 (.009) | .032 (.010) | .034 (.007)

7. Primary Outcome: Breath Alcohol Concentration (BrAC)
Description: Breath alcohol level will be measured using a breathalyzer repeatedly during the experimental session
Time Frame: Timepoint 7 (30 minutes after Timepoint 6)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
g/dL | .023 (.010) | .024 (.011) | .027 (.008)

8. Primary Outcome: Breath Alcohol Concentration (BrAC)
Description: Breath alcohol level will be measured using a breathalyzer repeatedly during the experimental session
Time Frame: Timepoint 8 (30 minutes after Timepoint 9)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
g/dL | .016 (.011) | .018 (.011) | .020 (.008)

9. Primary Outcome: Breath Alcohol Concentration (BrAC)
Description: Breath alcohol level will be measured using a breathalyzer repeatedly during the experimental session
Time Frame: Timepoint 9 (30 minutes after Timepoint 8)
Measure: Median (Standard Deviation); unit: g/dL
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 28 | 26 | 27
g/dL | .013 (.012) | .012 (.011) | .013 (.009)

10. Primary Outcome: Biphasic Effects of Alcohol (BAES)--Stimulation Subscale
Description: BAES stimulation will be measured by self-report repeatedly during the experimental session. The total score on the stimulation subscale ranges from 0-70 where higher is more stimulated.
Time Frame: Timepoint 1 (20 minutes after alcohol consumption is complete)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 9.40 (15.47) | 13.64 (20.01) | 14.07 (18.15)

11. Primary Outcome: Biphasic Effects of Alcohol (BAES)--Stimulation Subscale
Description: as for outcome 10
Time Frame: Timepoint 2 (30 minutes after Timepoint 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 26
score on a scale | 26.17 (17.54) | 27.82 (16.20) | 25.74 (16.27)

12. Primary Outcome: Biphasic Effects of Alcohol (BAES)--Stimulation Subscale
Description: as for outcome 10
Time Frame: Timepoint 3 (30 minutes after Timepoint 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 19.66 (15.24) | 21.39 (14.56) | 18.78 (15.01)

13. Primary Outcome: Biphasic Effects of Alcohol (BAES)--Stimulation Subscale
Description: as for outcome 10
Time Frame: Timepoint 4 (30 minutes after Timepoint 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 15.10 (14.33) | 14.14 (12.25) | 15.78 (14.73)

14. Primary Outcome: Biphasic Effects of Alcohol (BAES)--Stimulation Subscale
Description: as for outcome 10
Time Frame: Timepoint 5 (30 minutes after Timepoint 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 11.07 (12.18) | 11.96 (11.17) | 11.56 (13.00)

15. Primary Outcome: Biphasic Effects of Alcohol (BAES)--Stimulation Subscale
Description: as for outcome 10
Time Frame: Timepoint 6 (30 minutes after Timepoint 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 9.07 (9.86) | 8.18 (9.85) | 8.81 (11.94)

16. Primary Outcome: Biphasic Effects of Alcohol (BAES)--Stimulation Subscale
Description: as for outcome 10
Time Frame: Timepoint 7 (30 minutes after Timepoint 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 6.86 (9.60) | 6.68 (10.22) | 8.33 (12.04)

17. Primary Outcome: Biphasic Effects of Alcohol (BAES)--Stimulation Subscale
Description: as for outcome 10
Time Frame: Timepoint 8 (30 minutes after Timepoint 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 5.44 (8.27) | 5.81 (7.66) | 5.93 (8.53)

18. Primary Outcome: Biphasic Effects of Alcohol (BAES)--Stimulation Subscale
Description: as for outcome 10
Time Frame: Timepoint 9 (30 minutes after Timepoint 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 28 | 27 | 27
score on a scale | 4.96 (7.63) | 4.89 (7.55) | 6.78 (8.31)

19. Primary Outcome: Biphasic Effects of Alcohol--Sedation Subscale
Description: BAES sedation will be measured by self-report repeatedly during the experimental session. The total score on the sedation subscale ranges from 0-70 where higher is more sedated
Time Frame: Timepoint 1 (20 minutes after alcohol consumption is complete)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 2.66 (5.18) | 4.18 (6.06) | 3.78 (5.21)

20. Primary Outcome: Biphasic Effects of Alcohol--Sedation Subscale
Description: as for outcome 19
Time Frame: Timepoint 2 (30 minutes after Timepoint 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 12.31 (10.04) | 13.75 (10.66) | 11.81 (10.01)

21. Primary Outcome: Biphasic Effects of Alcohol--Sedation Subscale
Description: as for outcome 19
Time Frame: Timepoint 3 (30 minutes after Timepoint 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 15.45 (12.40) | 14.07 (11.31) | 13.41 (12.01)

22. Primary Outcome: Biphasic Effects of Alcohol--Sedation Subscale
Description: as for outcome 19
Time Frame: Timepoint 4 (30 minutes after Timepoint 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 15.76 (13.91) | 17.86 (14.41) | 14.15 (13.96)

23. Primary Outcome: Biphasic Effects of Alcohol--Sedation Subscale
Description: as for outcome 19
Time Frame: Timepoint 5 (30 minutes after Timepoint 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 15.41 (14.53) | 13.29 (12.36) | 12.89 (13.86)

24. Primary Outcome: Biphasic Effects of Alcohol--Sedation Subscale
Description: as for outcome 19
Time Frame: Timepoint 6 (30 minutes after Timepoint 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 14.86 (15.01) | 12.11 (13.14) | 12.00 (14.05)

25. Primary Outcome: Biphasic Effects of Alcohol--Sedation Subscale
Description: as for outcome 19
Time Frame: Timepoint 7 (30 minutes after Timepoint 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 11.72 (14.69) | 9.96 (11.30) | 10.48 (12.19)

26. Primary Outcome: Biphasic Effects of Alcohol--Sedation Subscale
Description: as for outcome 19
Time Frame: Timepoint 8 (30 minutes after Timepoint 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 8.31 (12.31) | 9.22 (10.78) | 8.74 (10.85)

27. Primary Outcome: Biphasic Effects of Alcohol--Sedation Subscale
Description: as for outcome 19
Time Frame: Timepoint 9 (30 minutes after Timepoint 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 28 | 27 | 27
score on a scale | 8.07 (10.86) | 6.70 (8.09) | 6.89 (7.90)

28. Primary Outcome: Alcohol Urge Questionnaire (AUQ
Description: The AUQ is a self-report measure of urge for alcohol and has been validated for real-time assessment of alcohol craving in the laboratory. The total score on the measure ranges from 0-48 where higher is worse
Time Frame: Timepoint 1 (20 minutes after alcohol consumption is complete)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 19.0 (7.95) | 19.82 (7.79) | 18.26 (8.19)

29. Primary Outcome: Alcohol Urge Questionnaire (AUQ
Description: as for outcome 28
Time Frame: Timepoint 2 (30 minutes after Timepoint 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 22.76 (10.52) | 23.14 (11.26) | 23.96 (10.51)

30. Primary Outcome: Alcohol Urge Questionnaire (AUQ
Description: as for outcome 28
Time Frame: Timepoint 3 (30 minutes after Timepoint 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 21.79 (9.42) | 21.25 (10.08) | 221.93 (10.08)

31. Primary Outcome: Alcohol Urge Questionnaire (AUQ
Description: as for outcome 28
Time Frame: Timepoint 4 (30 minutes after Timepoint 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 19.93 (8.38) | 19.21 (9.55) | 19.56 (8.73)

32. Primary Outcome: Alcohol Urge Questionnaire (AUQ
Description: as for outcome 28
Time Frame: Timepoint 5 (30 minutes after Timepoint 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 19.03 (7.76) | 18.46 (9.08) | 18.67 (8.50)

33. Primary Outcome: Alcohol Urge Questionnaire (AUQ
Description: as for outcome 28
Time Frame: Timepoint 6 (30 minutes after Timepoint 5)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 18.59 (8.67) | 19.21 (10.58) | 17.19 (7.77)

34. Primary Outcome: Alcohol Urge Questionnaire (AUQ
Description: as for outcome 28
Time Frame: Timepoint 7 (30 minutes after Timepoint 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 17.79 (7.89) | 17.54 (9.49) | 16.85 (7.61)

35. Primary Outcome: Alcohol Urge Questionnaire (AUQ
Description: as for outcome 28
Time Frame: Timepoint 8 (30 minutes after Timepoint 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on a scale | 16.83 (8.21) | 17.67 (10.51) | 16.11 (7.98)

36. Primary Outcome: Alcohol Urge Questionnaire (AUQ
Description: as for outcome 28
Time Frame: Timepoint 9 (30 minutes after Timepoint 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
Number analyzed (Participants) | 28 | 27 | 27
score on a scale | 17.04 (8.10) | 17.41 (9.78) | 15.59 (7.78)

ADVERSE EVENTS:
Time Frame: Participants were assessed during each study visit in related to baseline (for up to three study visits per participant), with each visit lasting 5 hours.
Arm/Group | 200mg Cannabidiol | 30mg Cannabidiol, | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT06105138/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT06105138/ICF_001.pdf